CLINICAL TRIAL: NCT00372320
Title: Open-Label, Dose-Escalation Study Evaluating the Safety of a Single Administration of AdhAQP1, an Adenoviral Vector Encoding Human Aquaporin-1 to One Parotid Salivary Gland in Individuals With Irradiation-Induced Parotid Salivary Hypofunction
Brief Title: Effect of AdhAQP1 on Salivary Flow in Patients Treated With Radiation for Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060206; 06-D-0206
Record Dates: First submitted 2006-09-02; First posted 2006-09-06 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09-05

CONDITIONS: Parotid Salivary Dysfunction
Keywords: Adenovirus; Aquaporin-1; Gene Transfer; Radiation-Induced Salivary Hypofunction; Salivary Gland; Xerostomia; Salivary Dysfunction; Hyposalivation; Dry mouth; head and neck cancer; side effects radiation damage
MeSH Terms: conditions — Adenoviridae Infections; Xerostomia; Head and Neck Neoplasms | interventions — Genetic Engineering

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Genetic: Gene Transfer
Drug: AdhAQP1

SUMMARY:
This study will examine whether the experimental drug AdhAQP1 can increase salivary flow in patients whose parotid glands have been exposed to therapeutic radiation for treatment of head and neck cancer. Radiation may damage the parotid glands (salivary glands located under the skin in front of the ear), leading to dry mouth, infections, excessive tooth decay, mouth sores, difficulty swallowing and pain. AdhAQP1 contains the human aquaporin-1 gene, which codes for a protein that works to transport water across cells, and a virus that normally can cause colds in humans, but is modified to render it ineffective. In animal experiments, AdhAQP1 has increased saliva production for a short time.

Patients between 18 years of age or older who received radiation treatment for head and neck cancer at least 5 years before enrolling in this study, who have no evidence of recurrent tumor, who have dry mouth and who secrete abnormally low levels of saliva from the parotid glands may be eligible for this study. Candidates are screened with a medical history, physical examination, blood, urine and saliva tests, electrocardiogram (EKG), chest x-ray, MRI exam, gallium scan (a nuclear medicine test to look for inflammation in the salivary glands), technetium pertechnetate scan (a nuclear medicine test to examine salivary gland function), parotid sialogram (x-ray of parotid gland), PET and CT scans to look for signs of tumor and a skin biopsy to collect skin cells for use in immunological tests.

Participants have a salt and sugar solution infused through a catheter (plastic tube) into both parotid glands. After 10 minutes, the solution drains into the mouth and is swallowed. Saliva is collected from the parotid glands at 6 and 24 hours after administration of the salt and sugar solution. Ten to 14 days later, patients are admitted to the NIH Clinical Center for up to 4 days for the following tests and procedures:

* On the first day, administration, through a catheter, of the study drug AdhAQP1 into one parotid gland.
* Monitoring over the next 3 days for changes in patients' ability to produce saliva. This includes medical examinations and several blood, urine and saliva collections.
* Technetium scan on day 2.
* Gallium scan on day 2.

Patients return to NIH for follow-up visits at 1, 2, 4, and 6 weeks after the AdhAQP1 infusion and then 3, 4, 5, 6 and 12 months for a medical examination and blood, urine and saliva collections. Gallium, technetium and MRI scans are repeated at several of the follow-up visits, and sialograms are done at 6 and 12 months. Chest x-ray and EKG are repeated at 4 and 6 months.

DETAILED DESCRIPTION:
The treatment of most head and neck cancer patients includes ionizing radiation (IR). Salivary glands in the IR field suffer irreversible damage. There is no conventional treatment available to correct this condition. Our research group has been developing the AdhAQP1 recombinant serotype 5 adenoviral (rAd5) vector based on the hypothesis that a replication deficient rAd5 vector is capable of safely transferring the human aquaporin-1 (hAQP1) cDNA to parotid glands of adult patients with IR-induced salivary hypofunction, resulting in an elevated salivary output, albeit transiently. Salivary glands have proven to be valuable gene transfer targets in numerous pre-clinical animal model studies. hAQP1, the archetypal water channel, is a plasma membrane protein that facilitates water movement across lipid bilayers. Rat and minipig studies have clearly shown that the AdhAQP1 strategy for restoring salivary flow to IR-damaged salivary glands is effective, and studies in rats, non-human primates and minipigs have shown that AdhAQP1 and similar rAd5 vectors are without significant untoward effects after salivary gland delivery. The purpose of this clinical protocol is to test the safety of AdhAQP1, with some measures of efficacy, in adult patients with established IR-induced parotid gland hypofunction. The targeted tissue site for the AdhAQP1 vector in the proposed study is a single parotid gland. In this Phase 1 dose-escalation study, safety will be evaluated using conventional clinical and immunological parameters. The primary outcome measure for biological efficacy will be parotid gland salivary output.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18 years of age or older.
  2. Capable of providing informed consent.
  3. History of radiation therapy for head and neck cancer, having received >45Gy to the parotid gland(s) due to primary or neck radiation.
  4. Abnormal parotid gland function in the targeted parotid gland as judged by absence of unstimulated parotid salivary flow and a stimulated parotid salivary flow in the targeted parotid gland <0.2 mL/min/gland after 2% citrate stimulation.
  5. Abnormal (99m)TcO4 scintiscan (reduced or absent uptake of (99m)TcO4) for the targeted parotid gland in the following circumstance: A (99m)TcO4 scintiscan will only be performed and used to determine eligibility if the isotope is available. If the isotope is not available, this inclusion criterion is not applicable.
  6. Abnormal sialogram (an altered ductal network with sialectasis) for the targeted parotid gland.
  7. No current evidence of malignancy by otolaryngology assessment, including a clinical history, nasopharyngolaryngoscopy, and negative CT or PET scan (e.g. reference 58).
  8. Absence of shedding wild type adenovirus in the saliva sample collected from the targeted gland at the pre-dose visit 1. Specifically, an aliquot of the pre-dose visit 1 saliva sample from the target parotid gland will be used to infect A549 cells to test for the presence of shedding WT Ad virus. If infectious virus emerges during the subsequent 7-10 day follow-up period, then the participant will no longer be eligible for treatment and will be withdrawn from the study. However, if no cytopathic effects are observed over a 7-10 day period, the participant may be treated provided all other eligibility criteria are met. If stimulated saliva cannot be collected at the pre-dose visit 1, this inclusion criterion is not applicable.
  9. Must be disease-free for at least 5 years, with the disease-free interval calculated from date of last cancer treatment (i.e., date of last radiation, chemotherapy or surgery) to date of pre-dose visit 1.
  10. Willingness to practice the required birth control method ("barrier" contraception, i.e., condoms, diaphragm) until AdhAQP1 is no longer detectable in their serum or saliva. Women who cannot bear children (post menopausal or due to a surgical intervention) also will be required to practice barrier birth control methods until AdhAQP1 is no longer detectable in their serum or saliva.
  11. Able to stay at the NIH hospital for the period of time necessary to complete each on-site phase of the protocol.
  12. No history of allergies to any medications or agents to be used in this protocol.
  13. On stable doses of medications (greater than or equal to 2 months from the pre-dose visit 1) for any underlying medical conditions.

EXCLUSION CRITERIA:

1. Pregnant or lactating women. Women of childbearing potential are required to have a negative serum pregnancy test at pre-dose visit 1 and a negative urine pregnancy test within 24 hours of treatment.
2. Any experimental therapy within 3 months of planned AdhAQP1 administration (Day 1).
3. Any active respiratory tract infection in the 3 weeks prior to planned AdhAQP1 administration (Day 1).
4. Active infection that requires the use of intravenous antibiotics and does not resolve at least 1 week before planned AdhAQP1 administration (Day 1).
5. Evidence of active substance or alcohol abuse or history of substance or alcohol abuse within two years of pre-dose visit 1.
6. Uncontrolled ischemic heart disease: unstable angina, evidence of active ischemic heart disease on ECG, congestive heart failure (left ventricular ejection fraction < 45% on MUGA or echo) or cardiomyopathy.
7. Asthma or chronic obstructive pulmonary disease requiring regular inhaled or systemic corticosteroids.
8. Individuals taking prescription medications (anti-cholinergics, anti-depressants) likely to result in salivary hypofunction.
9. Individuals with a history of autoimmune diseases affecting salivary glands, including Sj(SqrRoot)(Delta)gren s syndrome, lupus, scleroderma, type 1 diabetes, sarcoidosis, amyloidosis, and chronic graft versus host disease.
10. Use of systemic immunosuppressive medications, e.g., corticosteroids. Topical corticosteroids are allowed.
11. History of a second malignancy, within the past 3 years, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix.
12. Active hepatitis B, hepatitis C or HIV infection tested using blood collected at pre-dose visit 1.
13. WBC <3000/microL or ANC <1500/microL or Hgb <10.0 g/dL or platelets <100,000/microL or absolute lymphocyte count less than or equal to 500/microL using blood collected at pre-dose visit 2.
14. ALT and/or AST > 1.5 times the upper limit of normal (ULN) or alkaline phosphatase >1.5 times ULN using blood collected at pre-dose visit 2.
15. Serum creatinine > 2 mg/dL using blood collected at pre-dose visit 2.
16. Individuals who are active smokers.
17. Individuals who consume more than one alcoholic beverage/day.
18. Individuals who have an allergy to iodine or shellfish and thus are unable to have sialographic evaluations.
19. Individuals whose targeted parotid duct is not clinically accessible on screening sialography evaluations.
20. Individuals who on sialography have a distal stenosis in the targeted parotid gland that would impede vector delivery.
21. Individuals who likely would require use of a general anesthetic for ultrasound- guided core needle biopsy (applicable only for participants in dose cohorts 2-5).
22. Significant concurrent or recently diagnosed (<2 months from Day 1) medical condition that, in the opinion of the Medically Responsible Investigator, could affect the participant's ability to tolerate or complete the study.
23. Live vaccines within 4 weeks of first infusion.
24. Previous participation in a rAd5 vector gene transfer study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-09-01; Primary Completion 2014-03-19 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of single doses of escalating doses of AdhAQP1

SECONDARY OUTCOMES:
To evaluate the effectiveness of AdhAQP1 to increase parotid gland salivary output and improve symptoms associated with irradiation-induced parotid hypofunction.
To assess salivary flow in the treated parotid gland for up to three years.

CONTACTS AND LOCATIONS:
Overall Officials: Blake M Warner, D.D.S., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baum BJ, Wellner RB, Zheng C. Gene transfer to salivary glands. Int Rev Cytol. 2002;213:93-146. doi: 10.1016/s0074-7696(02)13013-0. PMID 11837896
- [Background] Zufferey R, Aebischer P. Salivary glands and gene therapy: the mouth waters. Gene Ther. 2004 Oct;11(19):1425-6. doi: 10.1038/sj.gt.3302321. No abstract available. PMID 15269715
- [Background] Baum BJ, Voutetakis A, Wang J. Salivary glands: novel target sites for gene therapeutics. Trends Mol Med. 2004 Dec;10(12):585-90. doi: 10.1016/j.molmed.2004.10.003. PMID 15567328
- [Derived] Alevizos I, Zheng C, Cotrim AP, Liu S, McCullagh L, Billings ME, Goldsmith CM, Tandon M, Helmerhorst EJ, Catalan MA, Danielides SJ, Perez P, Nikolov NP, Chiorini JA, Melvin JE, Oppenheim FG, Illei GG, Baum BJ. Late responses to adenoviral-mediated transfer of the aquaporin-1 gene for radiation-induced salivary hypofunction. Gene Ther. 2017 Mar;24(3):176-186. doi: 10.1038/gt.2016.87. Epub 2016 Dec 20. PMID 27996967
- [Derived] Baum BJ, Zheng C, Alevizos I, Cotrim AP, Liu S, McCullagh L, Goldsmith CM, McDermott N, Chiorini JA, Nikolov NP, Illei GG. Development of a gene transfer-based treatment for radiation-induced salivary hypofunction. Oral Oncol. 2010 Jan;46(1):4-8. doi: 10.1016/j.oraloncology.2009.09.004. Epub 2009 Nov 4. PMID 19892587